CLINICAL TRIAL: NCT00464971
Title: Evaluation of Safety and Efficacy of 17-Beta Estradiol in Treatment of Estrogen Deficiency-Derived Atrophic Vaginitis
Brief Title: Evaluation of Safety and Efficacy of 17-Beta Estradiol in Treatment of Atrophic Vaginitis: An Extension Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAG/PD/012/USA
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estradiol, 25 mcg

SUMMARY:
This trial was conducted in the United States of America (USA). This trial aimed to evaluate safety and efficacy of 17-beta Estradiol in the treatment of atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Postmenopausal
* Hysterectomized or non-hysterectomized
* Moderate or severe vaginal dryness and soreness
* Successful completion of the study VAG/PD/009/USA

Exclusion Criteria:

* Known, suspected, or past history of breast cancer
* Known, suspected, or past history of hormone-dependent tumor
* Genital bleeding of unknown etiology
* Acute thrombophlebitis or thromboembolic disorders or a past history of these conditions, associated with previous estrogen use
* Subjects who had adverse events during the final visit, or discontinued prematurely, or were noncompliant in VAG/PD/009/USA
* Exposure to any investigational new drug (other than what was dispensed in VAG/PD/009/USA) within the previous 30 days

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 1995-01-31 (Actual); Primary Completion 1996-11-30 (Actual); Study Completion 1996-11-30 (Actual)

PRIMARY OUTCOMES:
Relief of vaginal symptoms | over 12 months of treatment
Safety: Long-term effect on the endometrium assessed through evaluation of endometrial biopsies. AEs, clinical laboratory data and serum hormone levels

SECONDARY OUTCOMES:
Vaginal health, vaginal cytology and urethral cytology

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- [Derived] Bachmann G, Lobo RA, Gut R, Nachtigall L, Notelovitz M. Efficacy of low-dose estradiol vaginal tablets in the treatment of atrophic vaginitis: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):67-76. doi: 10.1097/01.AOG.0000296714.12226.0f. PMID 18165394
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com